CLINICAL TRIAL: NCT00918567
Title: Effects of Strattera and Behavior Therapy on the School and Home Functioning of Elementary School Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Impact of Strattera and Behavior Therapy on the Home and School Functioning of Children With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, James Waxmonsky, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B4Z-US-X053
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Atomoxetine; Behavior Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Drug Therapy; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined therapy (Experimental): atomoxetine plus behavior therapy
  Interventions: Drug: atomoxetine; Behavioral: Behavior Modification Therapy
- Drug therapy (Active Comparator): atomoxetine alone
  Interventions: Drug: atomoxetine

INTERVENTIONS:
Drug: atomoxetine — open label treatment dosed up to 1.8mg/kg/day
  Other Names: Drug Therapy
Behavioral: Behavior Modification Therapy — 8 week behavioral modification course with school consultation, parenting groups using COPE and child social skills group
  Other Names: Behavior Therapy
  Arms: Combined therapy

SUMMARY:
Background: Multiple studies have found Atomoxetine (Strattera) to be efficacious but there is only one published study specifically designed to evaluate its efficacy in school settings. In this 7 week placebo-controlled study, Atomoxetine (ATX) at mean dose of 1.3 mg/kg, significantly reduced teacher rated ADHD symptoms (Weiss et al., 2005). However, children are typically referred for treatment because of "real life" problems in functioning, not symptoms (Pelham, Fabiano, & Massetti, 2005). While ATX has been found to produce functional improvements at home, the Weiss study found limited results in this area at school.

Furthermore, almost no research has examined the effects of combining ATX and behavior therapy (BT). In the MTA, adding BT to stimulants improved teacher ratings of hyperactivity/impulsivity and increased the number of subjects reaching optimal response (Swanson et al., 2001). Therefore, it is possible that the addition of BT to ATX may improve functional performance in the classroom. The effects of combined therapy may be even larger for ATX as monotherapy with nonstimulants produces smaller effect sizes than with stimulants.

Objective: The primary objective was to evaluate the effects of ATX alone and in combination with BT on the school functioning of 56 children ages 6-12 with ADHD. Outcomes were assessed using traditional symptoms measures as well as functional measures of academic and behavioral improvements in the classroom.

DETAILED DESCRIPTION:
The objectives were evaluated in an 8 week open label trial of where half of the participants were randomly assigned to receive (ATX+BT) while the rest received only ATX. An open label design was employed as the efficacy of ATX for ADHD symptoms has been established and to ensure that all patients received at least one active treatment. Parents in the ATX+BT group attended an eight week parenting course using the Community Oriented Parent Education (COPE) program (Cunningham, Bremner, & Secord, 1998) while the child participated in an eight week social skills course. Teachers implemented a Daily Report Card (DRC) to track classroom behaviors. In the BT group, the child's DRC performance was communicated daily to parents and tied to consequences at home and school. In the ATX group, parents were not provided with the DRCs. The ATX dosing protocol was as follows: .5mg/kg per day on days 1-3, .8mg/kg/day days 4-7, 1.2mg/kg days 8+. After 3 weeks, subjects were eligible to increase to 1.8mg/kg/day. ATX was dosed once in the morning but could be dosed BID to address tolerability. The mean final dose was 1.4mg/kg/day.

To be enrolled, children must have had an IQ > 75, not failed a trial of ATX, met DSM criteria for ADHD but not other psychiatric comorbidities except ODD/CD and be in good physical health. Children already taking ADHD medication were enrolled only if the average symptom score on the ADHD subscale of the Disruptive Behaviors Disorders (DBD) scale was >2 (moderate impairment). ADHD was confirmed by parent report on the DISC and the DBD, which rates all DSM 3R and IV symptoms of ODD, CD and ODD on a 0-3 likert scale. Subjects were also required to evidence ADHD symptoms in the classroom as rated on the IOWA Conners. Psychiatric comorbidities were assessed using the DISC.

Measures of treatment response included:

1. Parents and teacher ratings on the IOWA Conners: 10 item Likert ratings to measure children's inattention-overactive-impulsive and oppositional-defiant behavior (Milich, Loney, & Landau, 1982)
2. Parent and teacher ratings on the Impairment Rating Scale (IRS): 8 items using visual-analogue scales to measure children's functional impairment in peer relationships, adult-child relationships, academic performance, classroom behavior, and self esteem (Fabiano et al., 2006).
3. Parent and teacher side effect ratings using a structured list of common side effects seen with ATX modeled after the Pittsburgh Side Effects Rating Scale (Pelham, 1993).
4. Direct observations of subjects to measure rule violations and on/off task behavior using a modified version of the COCADD system (Atkins, Pelham & Licht, 1988) in which trained observers watched children in their classroom for 30 minutes, recording each rule violation and off-task behavior.
5. Parent and teacher rating on the Social Skills Rating Scale (SSRS): a measure of teachers' and parents perceptions of children's social and academic skills and of their overall problem behaviors (Gresham & Elliott, 1990).

ELIGIBILITY:
Inclusion Criteria:

1. meet DSM-IV diagnostic criteria for ADHD-combined type;
2. estimated IQ of 75 or higher;
3. agree to comply with the randomly assigned treatment condition;
4. enrolled in full time school at first grade level or higher; AND
5. have a primary teacher available to complete ratings for the entire study duration.

Exclusion Criteria:

1. current or past history of seizures (not including benign febrile seizures) or other neurological disorders;
2. physical conditions that preclude administration of Strattera or other medical illness that might confound study results or increase the safety risk to subjects exposed to study treatments (i.e. marked cardiac conduction delay, etc.);
3. prior failed trial of Strattera defined as 3 weeks or more on a daily dose of Strattera of at least .8mg/kg or a documented inability to tolerate at least .8mg/kg/day;
4. serious forms of psychopathology other than ADHD, such autism, bipolar disorder, schizophrenia or any other psychopathology requiring urgent treatment with psychotropic medication; OR
5. children for whom discontinuation of their current psychotropic medication would represent a serious risk to themselves or others.

The presence of Oppositional Defiant Disorder (ODD), Conduct Disorder (CD) or learning disabilities will not result in exclusion from the study as they are commonly occurring comorbidities that have not been found to moderate response to ADHD treatments (Jensen et al., 2001). Enrollment in special education services will also not be an exclusionary criteria as work by this research group has found that such services do not affect response to ADHD treatments (Niemic, Fabiano, Pelham, & Fuller, 2002).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James G Waxmonsky, Principal Investigator — SUNY Buffalo; Daniel A Waschbusch, Principal Investigator — SUNY Buffalo
Locations (1):
- Cennter for Children and Families, Buffalo, New York, United States

REFERENCES:
- [Derived] Waxmonsky JG, Waschbusch DA, Pelham WE, Draganac-Cardona L, Rotella B, Ryan L. Effects of atomoxetine with and without behavior therapy on the school and home functioning of children with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2010 Nov;71(11):1535-51. doi: 10.4088/JCP.09m05496pur. Epub 2010 Jun 29. PMID 20673557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from schools, pediatric offices and the local community through radio and print advertisement. Subjects were recruited between Jan of 2007 and the spring of 2008.
Pre-assignment Details: uneven number because set of twins randomized as one unit at parental request
Period: Overall Study
Arm/Group | Combined Therapy | Drug Therapy
Started | 29 | 27
Completed | 24 | 25
Not Completed | 5 | 2
Not completed — Lack of Efficacy | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Therapy | Drug Therapy | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 27 | 56
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (1.6) | 8.9 (1.5) | 8.59 (1.581)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Rule Violations During Direct Classroom Observation at Endpoint (Week 8)
Description: Observations were conducted using the Student Behavior Teacher Response Observation Code. After learning the classroom rules, observers watched children in their classrooms for 30 minutes during an academic activity and recorded each time the subject violated a classroom rule. Total classroom rule violations were used as the primary outcome measures for the study.
Time Frame: Endpoint (Week 8)
Population: all subjects analyzed using ITT
Measure: Mean (Standard Error); unit: number occurences per 30 mins
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
number occurences per 30 mins | 6.15 (1.37) | 4.93 (1.36)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also tested marginal effects defined as p < .10; Tukey-Kramer adjustments for post-hoc differences of least squares comparisons; Mean Difference (Final Values) = -1.22, Standard Error of Mean 1.93

2. Secondary Outcome: Impairment Rating Scale (Parent Completed) at Endpoint
Description: The IRS is a 8 item measure that uses visual-analogue scales to evaluate the child's problem level and need for treatment in developmentally important areas, such as peer relationships, adult-child relationships, academic performance, and classroom behavior 51. The scale is scored from 0 (no problem) to 6 (extreme problem). The scale has excellent test-retest and inter-rater reliability and well supported validity 51, 52.
Time Frame: Endpoint (Week 8)
Population: Intent to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | 2.66 (.37) | 2.84 (.36)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also examined marginal effects, defined as p<.10; Mean Difference (Final Values) = 0.18, Standard Error of Mean 0.51

3. Secondary Outcome: Impairment Rating Scale (Teachers) at Endpoint
Description: The IRS is a 6 item measure that uses visual-analogue scales to evaluate the child's problem level and need for treatment in developmentally important areas, such as peer relationships, adult-child relationships, academic performance, and classroom behavior. The scale is scored from 0 (no problem) to 6 (extreme problem). The scale has excellent test-retest and inter-rater reliability and well supported validity.
Time Frame: Endpoint (Week 8)
Population: ITT was used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | 2.02 (0.42) | 2.29 (0.43)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also tested marginal effects defined as p<.10; Mean Difference (Final Values) = 0.27, Standard Error of Mean 0.60

4. Secondary Outcome: Pittsburgh Side Effects Rating Scale (PSERS)(Parent Completed) at Endpoint:
Description: The PSERS measures adverse events commonly associated with stimulant medication and has been used in multiple studies of ADHD. For this study, the PSERS was modified to also assess adverse emotional events potentially associated with ATX, including suicidal statements. The resulting scale consisted of 14 items (an additional sleep item for parents) rated from 0 ("none") to 3 ("severe"). An overall side effects score was computed by averaging across all ratings and used in analyses.
Time Frame: Endpoint (Week 8)
Population: ITT was used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | .38 (.06) | .34 (.06)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also estimated marginal effects defined as p<.10; Mean Difference (Final Values) = -0.05, Standard Error of Mean 0.09

5. Secondary Outcome: Pittsburgh Side Effects Rating Scale (PSERS)(Teacher Rated):
Description: The PSERS measures adverse events commonly associated with stimulant medication and has been used in multiple studies of ADHD. For this study, the PSERS was modified to also assess adverse emotional events potentially associated with ATX, including suicidal statements. The resulting scale consisted of 13 items (for teachers) rated from 0 ("none") to 3 ("severe"). An overall side effects score was computed by averaging across all ratings and used in analyses.
Time Frame: at weeks 8 (Endpoint)
Population: ITT was used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | .23 (.05) | .21 (.05)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — also tested marginal effects defined as p<.10; Mean Difference (Final Values) = -0.02, Standard Error of Mean 0.07

6. Secondary Outcome: Disruptive Behavior Disorders Rating Scale ODD Subscale (DBD- Parent Completed) at Endpoint
Description: The DBD consists of 8 items that are the DSM-IV symptoms of Oppositional Defiant Disorder (ODD). Items on the DBD were rated by parents and teachers using Likert scales that ranged from 0 ("not at all") to 3 ("very much"). The factor structure, reliability and validity of the DBD have been supported in multiple studies.
Time Frame: Endpoint (Week 8)
Population: ITT was used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | .90 (.13) | 1.12 (.13)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p > .05, Mixed Models Analysis — Also tested marginal effects defined as p<.10; Mean Difference (Final Values) = 0.22, Standard Error of Mean 0.18

7. Secondary Outcome: Disruptive Behavior Disorder Rating Scale ODD Subscale(DBD- Teacher Completed) at Endpoint
Description: as for outcome 6
Time Frame: Endpoint (Week 8)
Population: ITT was used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | .54 (.15) | .71 (.14)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also tested marginal effects (p<.10); Mean Difference (Final Values) = 0.17, Standard Error of Mean 0.20

8. Secondary Outcome: Social Skills Rating Scale Problem Behavior Subscale(SSRS Parent) at Endpoint
Description: completed by parents to measure children's problem behaviors (PB). Items are rated from 0 ("not at all") to 2 ("very often"). The scale has 55 items. The score reported below is the sum total of the items on the scale and then averaged for the whole group. Therefore, the range can be between 0 and 110. A higher score indicates a better outcome.
Time Frame: Endpoint (Week 8)
Population: ITT was used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | 16.48 (1.21) | 19.53 (1.19)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — Also tested marginal effects (p<.10); Mean Difference (Final Values) = 3.05, Standard Error of Mean 1.70

9. Secondary Outcome: Social Skills Rating Scale Problem Behavior Subscale(SSRS Teachers) at Endpoint
Description: The SSRS was completed by teachers to measure children's problem behaviors (PB). Items are rated from 0 ("not at all") to 2 ("very often"). The scale has 55 items. The score reported below is the sum total of the items on the scale and then averaged for the whole group. Therefore, the range can be between 0 and 110. A higher score indicates a better outcome.
Time Frame: Endpoint (Week 8)
Population: ITT was used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | 13.88 (1.25) | 13.96 (1.29)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also tested marginal effects (p<.10); Mean Difference (Final Values) = 0.08, Standard Error of Mean 1.80

10. Secondary Outcome: ADHD Subscale of the DBD (Parent Completed) at Endpoint
Description: The DBD consists of 18 items that are the DSM-IV symptoms of ADHD. Items on the DBD were rated by parents and teachers using Likert scales that ranged from 0 ("not at all") to 3 ("very much"). The factor structure, reliability and validity of the DBD have been supported in multiple studies.
Time Frame: Endpoint (Week 8)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | 1.07 (0.11) | 1.47 (0.11)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also tested marginal effect (p<.10); Mean Difference (Final Values) = 0.40, Standard Error of Mean 0.15

11. Secondary Outcome: ADHD Subscale of the DBD (Teacher Completed) at Endpoint
Description: The ADHD subscale of the DBD consists of 18 items that are the DSM-IV symptoms of ADHD. Items on the DBD were rated by parents and teachers using Likert scales that ranged from 0 ("not at all") to 3 ("very much"). The factor structure, reliability and validity of the DBD have been supported in multiple studies.
Time Frame: Endpoint (Week 8)
Population: ITT used
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Therapy | Drug Therapy
Number analyzed (Participants) | 29 | 27
units on a scale | 1.01 (0.13) | 1.13 (0.13)
Statistical Analysis 1: Comparison: Combined Therapy vs Drug Therapy; Test type: Superiority or Other; p < .05, Mixed Models Analysis — Also tested marginal effects (p<.10); Mean Difference (Final Values) = 0.12, Standard Error of Mean 0.19

ADVERSE EVENTS:
Time Frame: The Pittsburgh Side Effect Rating Scale (PSERS) measures adverse events commonly associated with ADHD medication rated from 0 ("none") to 3 ("severe"). Both teachers and parents completed it at weeks 1, 3 and 8.
Description: Because of concerns over adverse emotional reactions with three specific items were examined separate from the total score: (1) suicidal statements (e.g., "I wish I was dead"); (2) crabby/irritable; and (3) tearful, sad, depressed. In addition, weight, height and resting blood pressure were monitored at each office visit (weeks 0, 3 and 8).
Arm/Group | Combined Therapy | Drug Therapy
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 25/29 | 24/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Combined Therapy (N=29) | Drug Therapy (N=27)
Trouble Sleeping (Psychiatric disorders) | 4 (6) | 3 (4) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
stomachaches (Gastrointestinal disorders) | 8 (10) | 4 (7) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
appetite loss (Metabolism and nutrition disorders) | 7 (11) | 2 (4) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
headaches (Nervous system disorders) | 5 (6) | 3 (5) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
motor tics (Nervous system disorders) | 4 (7) | 4/7 (7) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
picking at skin (Psychiatric disorders) | 9 (16) | 10 (17) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
anxiety (Psychiatric disorders) | 10 (18) | 12 (14) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
dulled/tired looking (Psychiatric disorders) | 13 (15) | 10 (11) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
crabby/irritable (Psychiatric disorders) | 14 (19) | 11 (16) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8
depressed mood/crying episodes (Psychiatric disorders) | 8 (12) | 5 (6) — computed from PSERS ratings from parents & teachers at weeks 1,3+8; there were 2 cases (1 per group)of expressed suicidal ideation; these 2 subjects were assessed by study doctors; neither were found to have a genuine desire to commit suicide.
withdrawn from others (Psychiatric disorders) | 5 (10) | 3 (5) — computed from combined PSESR ratings from parents and teachers at weeks 1, 3 and 8

LIMITATIONS AND CAVEATS:
The primary limitation of this study was the lack of a control condition, thereby limiting our ability to detect the causality of observed improvements. Study may not have had sufficient subjects to detect group differences on secondary measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No